CLINICAL TRIAL: NCT01322880
Title: Microfinance-Discussion Session Intervention in Post-Conflict Central African States
Brief Title: Domestic Violence Discussion Session
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Economics and Political Science (Other)
Responsible Party: Radha Iyengar, London School of Economics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HF15660-101
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2009-02

CONDITIONS: Intimate Partner Violence
Keywords: domestic violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Other): The project, administered by the International Rescue Committee (IRC), involved 25 village savings and loans association (VSLA) groups across the province. The VSLA groups initially formed through local members of the community designated as community based facilitators (CBF).
  Interventions: Behavioral: Village Savings and Loans Associations
- Treatment Group (Experimental): Half of the VSLA participants were invited to participate in an additional set of discussion groups to be attended along with their spouse. All participants were informed that due to space constraints, only half of the members would be able to attend. In each VSLA, individuals drew numbers from a bag or hat, and those with "winning" slips were the ones who entered the discussion groups with spouses.
  Interventions: Behavioral: Discussion sessions; Behavioral: Village Savings and Loans Associations

INTERVENTIONS:
Behavioral: Discussion sessions — Those selected were invited to attend a 6 session course on household decision-making with their spouses. Topics included budgeting, household financial management, and negotiation skills
  Other Names: Household Financial Training
  Arms: Treatment Group
Behavioral: Village Savings and Loans Associations — The approach developed by CARE International develops Village Savings and Loan Associations (VSLAs). A VSLA is a self-selected group of people who pool their money into a fund from which members can borrow. The money is paid back with interest, causing the fund to grow. The regular savings contributions to the Association are deposited with an end date in mind for distribution of all or part of the total funds (including interest earnings) to the individual members, usually on the basis of a formula that links payout to the amount saved. This lump sum distribution provides a large amount of money that members can then use as they want, without restriction.
  Other Names: Village Microfinance

SUMMARY:
Over the last twenty years micro-finance based interventions have proven to be a popular and often effective means of improving the economic outcomes of impoverished women. However, the gains to microfinance based interventions on women's decision making in both economic and non-economic arenas remains largely unknown. Specifically, the question of to what extent does access to small-scale credit alone, rather than other programs often combined with microfinance, affect women's empowerment is of particular interest when determining interventions in a variety of setting in developing nations. There exists evidence that women's empowerment is associated with reduced violence and as such maybe an important tool for improving adult women's wellbeing. In addition increased decision making power by women has been associated with improvement in children's health outcomes, especially for girls, and as such may be way generating intergenerational improvements in women's outcomes.

The goal of this project is to disentangle the effects of access to credit alone from the information on financial and personal decision making that is frequently coupled with these programs. To accomplish this, the investigators use a randomized field experiment among participants in Village Savings and Loans Associations (VSLA's). VSLA participants are a self-selected group of people who pool their money into a fund from which members can borrow. The money is paid back with interest, causing the fund to grow. The regular savings contributions to the VSLA are deposited with an end date (usually less than 1 year) after which all or part of the total funds are distributed to the individual members. The small loans are paid back with interest which is determined by the group at the time of formation and the returns from these interest payments are also distributed to the groups. The investigators then test whether there are additional gains to women's well-being by providing VSLA participants with training on process-based decision making to determine if there is a need for additional efforts to improve the decision making structure in households. To the extent that increased access to credit and more broadly financial resources is limited by existing constraints on women's decision making power, this additional training may be a necessary part of the creation of credit markets in improving the health and well-being of women and children.

DETAILED DESCRIPTION:
* How are subjects recruited? What inducement is offered? If participants are paid, what amount and when are they paid? Is there partial pay for partial completion? (Append copy of letter or advertisement or poster, if any.)

Subjects are voluntary participants in a Village and Savings Group organized by the International Rescue Committee

* Salient characteristics of subjects--number who will participate, age range, sex, institutional affiliation, other special inclusion and exclusion criteria (if children, prisoners or other vulnerable subjects are recruited, explain why their inclusion is necessary):

Subjects will be 600 individuals, predominantly women, aged 20-50, who reside in the Burundi province of Makamba (in the southern part of Burundi)

* Describe how permission has been obtained from cooperating institution(s)--school, hospital, corporation, prison, or other relevant organization. (Append letters.) Is the approval of other research compliance committees or another Institutional Review Board required?

Jodi Nelson: (protocols)

* What do subjects do, or what is done to them, or what information is gathered? (Append copies of instructions, tests, questionnaires, or interview guides to be used.) How many times will observations, tests, etc., be conducted? How long will their participation take? Are interviews to be tape recorded or videotaped?

Everyone in the sample (N=600) is in a VSLA with its financial design previously determined. Half of the sample will be treated as the "control" group and will not receive the treatment. Of this sample, in half of the VSLA's the investigators will ask the spouse to accompany the member to one payment meeting. A baseline survey will be conducted in January 2008 to gather basic demographic information as well as pre-treatment levels of variables of interest The training/discussion groups will take place over several months are intended to promote joint decision-making. conduct a post-treatment survey to determine immediate gains from the treatment. After another 1-2 months, the investigators will conduct a final survey to determine the survival rate of any changes. Interviews will be recorded in written form to be input into computerized data management systems.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Village Savings and Loans Association program administered by International Rescue Committee--Burundi

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Domestic Violence Exposure | baseline, 6 months, 12 months, 15 months
  The measure of exposure to violence used in this survey is the Hurt Insult Threaten Scream (HITS) instrument. It includes four items: physical abuse, insults, threats and screaming. The four items are scored on a Likert 5-point scale. The HITS was chosen due to its proven applicability in a variety of settings , and because it allows for a rapid appraisal of past experiences of violence. Its measurement regards the two weeks prior to the interview. Similar to the more commonly used World Health Organization methodology, but includes indicators of abuse such as threats and insults.

SECONDARY OUTCOMES:
Attitudes towards gender roles and rights | Baseline, 6 months, 15 months
  Attitudinal questions on traditional gender roles and appropriateness of abuse in a range of common settings. The questions are based on those asked in the Demographic Health Survey funded by USAID
Economic Empowerment | baseline, 6 months, 12 months, 15 months
  The intervention aimed to improve decision making dynamics in this direction, encouraging both men and women to take increasingly more decisions jointly. We identified several areas which may be critical to women's empowerment: income/asset-related decision making authority, fertility decision making authority, safety, and legal and political rights

CONTACTS AND LOCATIONS:
Overall Officials: Radha Iyengar, PhD, Principal Investigator — London School of Economics and Political Science
Locations (1):
- International Rescue Committee--Burundi, Makamba, Makamba Province, Burundi

REFERENCES:
- See also: Supplementary Material for Intervention (training, survey instruments, instructions) — http://personal.lse.ac.uk/iyengarr/burundi_ipv.htm